CLINICAL TRIAL: NCT00427895
Title: A Phase 3, Randomized, Active-controlled, Modified Double-blind Trial Evaluating The Safety, Tolerability, And Immunogenicity Of A 13-valent Pneumococcal Conjugate Vaccine (13vpnc) Compared To A 23-valent Pneumococcal Polysaccharide Vaccine (23vps) In Adults 60 To 64 Years Old Who Are Naive To 23vps And The Safety, Tolerability, And Immunogenicity Of 13vpnc In Adults 18-59 Years Old Who Are Naïve To 23vps
Brief Title: Study Comparing a 13-valent Pneumococcal Conjugate Vaccine With 23-valent Pneumococcal Polysaccharide Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6115A1-004; B1851019 (Other: Alias Study Number); NCT00488852 (obsolete NCT alias); NCT00774410 (obsolete NCT alias)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Pneumococcal Infections
Keywords: Vaccine; Pneumococcal Infections Prevention and Control
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 13vPnC Cohort 1, Vaccination 1 (Experimental): Participants aged 60-64 years were given a 0.5 mL dose administered on day 1.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)
- 23vPS Cohort 1, Vaccination 1 (Active Comparator): Participants aged 60-64 years were given a 0.5 mL dose administered on day 1.
  Interventions: Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS)
- 13vPnC Cohort 2, Vaccination 1 (Experimental): Participants aged 50-59 years given a 0.5 mL dose administered on day 1.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)
- 13vPnC Cohort 3, Vaccination 1 (Experimental): Participants aged 18-49 years given a 0.5 mL dose administered on day 1.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)
- 13vPnC Cohort 1, Vaccination 2 (Experimental): Participants aged 60-64 years who received 13vPnC at vaccination 1 receive a 0.5 mL dose of 13vPnC administered 3-4 years after dose 1.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)
- 23vPS Cohort 1, Vaccination 2 (Active Comparator): Participants aged 60-64 years who received 23vPS at vaccination 1 receive a 0.5 mL dose of 23vPS administered 3-4 years after dose 1.
  Interventions: Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS)
- 13vPnC Cohort 2, Vaccination 2 (Experimental): Participants aged 50-59 years who received 13vPnC at vaccination 1 receive a 0.5 mL dose of 13vPnC administered 3-4 years after dose 1.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL dose administered on day 1
  Arms: 13vPnC Cohort 1, Vaccination 1
Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS) — 0.5 mL dose administered on day 1
  Arms: 23vPS Cohort 1, Vaccination 1
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL dose administered on day 1
  Arms: 13vPnC Cohort 2, Vaccination 1
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL dose administered on day 1
  Arms: 13vPnC Cohort 3, Vaccination 1
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL dose administered 3-4 years after dose 1
  Arms: 13vPnC Cohort 1, Vaccination 2
Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS) — 0.5 mL dose administered 3-4 years after dose 1
  Arms: 23vPS Cohort 1, Vaccination 2
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL dose administered 3-4 years after dose 1
  Arms: 13vPnC Cohort 2, Vaccination 2

SUMMARY:
This study will assess the safety, tolerability and immune response of 13-valent pneumococcal conjugate vaccine (13vPnC) compared with 23-valent Pneumococcal Polysaccharide Vaccine (23vPS). Although the study started with only 1 population, amendments to the original protocol will now reflect three participant populations. Three age cohorts will be enrolled. The first cohort (age 60-64) will be blinded. Cohort 2 (age 50-59) and cohort 3 (age 18-49) are open label. Subjects in cohorts 1 and 2 will receive 2 vaccinations 3-4 years apart. Subjects in cohort 3 will receive 1 vaccination. All participants should be naïve of 23vPS. Comparisons of immune responses from the different cohorts will be done.

ELIGIBILITY:
Inclusion Criteria:

* First Cohort: Healthy Male and female adults 60 to 64 years of age at time of enrollment.
* Second Cohort: Healthy Male and female adults 50 to 59 years of age at time of enrollment.
* Third Cohort: Healthy Male and female adults 18 to 49 years of age at time of enrollment.

Exclusion Criteria:

* Previous immunization with any licensed or experimental pneumococcal vaccine.
* Serious chronic disorders including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder which in the investigator's opinion precludes the subject from participating in the study.
* Known or suspected impairment of immunological function.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2141 (Actual)
Dates: Start 2007-02-27 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (25):
  - Accelovance, Huntsville, Alabama
  - East Valley Family Physicians, PLC, Chandler, Arizona
  - Clinical Research Advantage/Central Phoenix, Phoenix, Arizona
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Accelovance, South Bend, Indiana
  - Heartland Research Associates LLC, Wichita, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric /Adult Research, Bardstown, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research - St. Louis, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - PMG Research of Raleigh, LLC, Cary, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Primary Physicians Research, Upper Saint Clair, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Internal Medicine and Pediatrics Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristoll, LLC, Bristol, Tennessee
  - J. Lewis Research Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - J. Lewis Research/First Med, West Jordan, Utah
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-004&StudyName=Study%20Comparing%20a%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20With%2023-valent%20Pneumococcal%20Polysaccharide%20Vaccine%20in%20Adults

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Cohort 1 and 2 participated for 1 year in the study. Vaccination 2 (3 to 4 years after vaccination 1) was administered to participants in Cohort 1 and 2. Participants in Cohort 3 enrolled as part of amendment 3 participated for 6 months and participants in Cohort 3 enrolled as part of amendment 4 participated for 1 year in study.
Groups:
- 13vPnC, Cohort 1: Participants 60-64 years of age received 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a 0.5 milliliter (mL) single dose intramuscularly (Vaccination 1 [Vax1]) at baseline.
- 23vPS, Cohort 1: Participants 60-64 years of age received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose intramuscularly (Vaccination 1) at baseline.
- 13vPnC, Cohort 2: Participants 50-59 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly at (Vaccination 1) at baseline.
- 13vPnC, Cohort 3: Participants 18-49 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly (Vaccination 1) at baseline.
- 13vPnC/13vPnC, Cohort 1: Participants 60-64 years of age who received 13vPnC at vaccination 1, received open-label 0.5 mL single dose intramuscularly of 13vPnC (Vaccination 2) at Year 3 to 4.
- 13vPnC/23vPS, Cohort 1: Participants 60-64 years of age who received 13vPnC at vaccination 1, received open-label 0.5 mL single dose intramuscularly of 23vPS (Vaccination 2) at Year 3 to 4.
- 23vPS/23vPS, Cohort 1: Participants 60-64 years of age who received 23vPS at vaccination 1, received open-label 0.5 mL single dose intramuscularly of 23vPS (Vaccination 2) at Year 3 to 4.
- 13vPnC/13vPnC, Cohort 2: Participants 50-59 years of age who received 13vPnC at vaccination 1, received open-label 0.5 mL single dose intramuscularly of 13vPnC (Vaccination 2) at Year 3 to 4.
Period: Between 6-Month Follow-up - Year 1
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Started | 411 | 411 | 392 | 854 | 0 | 0 | 0 | 0
Completed | 411 | 411 | 392 | 502 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 352 | 0 | 0 | 0 | 0
Not completed — Did not enter 1-year blood draw | 0 | 0 | 0 | 352 | 0 | 0 | 0 | 0
Period: Vax 2/Year 3 to 4
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Started | 0 | 0 | 0 | 0 | 108 | 108 | 189 | 214
Completed | 0 | 0 | 0 | 0 | 107 | 108 | 189 | 212
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Failed to Return | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Vax 1 Baseline/6-Month Follow-up
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Started | 418 | 417 | 406 | 900 | 0 | 0 | 0 | 0
Vaccinated | 417 | 414 | 404 | 899 | 0 | 0 | 0 | 0
Completed | 411 | 411 | 392 | 854 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 14 | 46 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 4 | 32 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 7 | 0 | 0 | 0 | 0
Not completed — Failed to Return | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Randomized, Not Vaccinated | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Period: Vax 1/Year 1 Follow-up
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Started | 411 | 411 | 392 | 502 | 0 | 0 | 0 | 0
Completed | 404 | 396 | 373 | 469 | 0 | 0 | 0 | 0
Not Completed | 7 | 15 | 19 | 33 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 2 | 21 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 6 | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to Return | 0 | 0 | 12 | 5 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Between Year 1 - Vax 2/Year 3 to 4
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Started | 404 | 396 | 373 | 469 | 0 | 0 | 0 | 0
Completed | 216 | 189 | 214 | 0 | 0 | 0 | 0 | 0
Not Completed | 188 | 207 | 159 | 469 | 0 | 0 | 0 | 0
Not completed — Did Not Consent to Receive Vax 2 | 188 | 207 | 159 | 469 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC, Cohort 1: Participants 60-64 years of age received 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a 0.5 milliliter (mL) single dose intramuscularly (Vaccination 1 [Vax1]).
- 23vPS, Cohort 1: Participants aged 60-64 years old received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose intramuscularly (Vaccination 1).
- 13vPnC, Cohort 2: Participants 50-59 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly (Vaccination 1).
- 13vPnC, Cohort 3: Participants 18-49 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly (Vaccination 1).
- Total: Total of all reporting groups
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3 | Total
Number analyzed (Participants) | 417 | 414 | 403 | 899 | 2133
Age, Customized [Number; unit: participants] — In 13vPnc, Cohort 2; out of 404 participants vaccinated, 1 participant randomized and vaccinated in error without a consent form, and hence baseline characteristics are available for 403 participant.
  participants
    18 to 29 years | 0 | 0 | 0 | 300 | 300
    30 to 39 years | 0 | 0 | 0 | 298 | 298
    40 to 49 years | 0 | 0 | 0 | 301 | 301
    50 to 59 years | 0 | 0 | 403 | 0 | 403
    60 to 64 years | 417 | 414 | 0 | 0 | 831
Sex: Female, Male [Count of Participants; unit: Participants] — In 13vPnc, Cohort 2; out of 404 participants vaccinated, 1 participant randomized and vaccinated in error without a consent form, and hence baseline characteristics are available for 403 participant.
  Participants
    Female | 223 | 252 | 249 | 523 | 1247
    Male | 194 | 162 | 154 | 376 | 886

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 2 (Year 3 to 4) in Cohort 1 and Cohort 2
Description: Local reactions reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 cm; Moderate (5.1 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating); Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move arm above head; able to move arm above shoulder); Severe (unable to move arm above shoulder).
Time Frame: Within 14 days after vaccination 2
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants with known values for any local reaction. 'n'=number of participants with known values for specified local reaction for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 13vPnC/13vPnC, Cohort 1: Participants 60-64 years of age who received 13vPnC at vaccination 1, received a 0.5 mL single dose intramuscularly of open-label 13vPnC (Vaccination 2 [Vax2]) at Year 3 to 4.
- 23vPS/23vPS, Cohort 1: Participants aged 60-64 years of age who received 23vPS at vaccination 1, received a 0.5 mL single dose intramuscularly of open-label 23vPS (Vaccination 2) at Year 3 to 4.
- 13vPnC/23vPS, Cohort 1: Participants 60-64 years of age who received 13vPnC at vaccination 1, received a 0.5 mL single dose intramuscularly of open-label 23vPS (Vaccination 2) at Year 3 to 4.
- 13vPnC/13vPnC, Cohort 2: Participants 50-59 years of age who received 13vPnC at vaccination 1 received a 0.5 mL single dose intramuscularly of open-label 13vPnC (Vaccination 2) at Year 3 to 4.
Arm/Group | 13vPnC/13vPnC, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Number analyzed (Participants) | 80 | 167 | 89 | 174
Percentage of participants
  Redness: Any: number analyzed (Participants) | 50 | 109 | 51 | 84
  Redness: Any | 20.0 [10.0 to 33.7] | 35.8 [26.8 to 45.5] | 27.5 [15.9 to 41.7] | 21.4 [13.2 to 31.7]
  Redness: Mild: number analyzed (Participants) | 50 | 101 | 49 | 83
  Redness: Mild | 20.0 [10.0 to 33.7] | 27.7 [19.3 to 37.5] | 22.4 [11.8 to 36.6] | 18.1 [10.5 to 28.0]
  Redness: Moderate: number analyzed (Participants) | 48 | 91 | 44 | 75
  Redness: Moderate | 6.3 [1.3 to 17.2] | 18.7 [11.3 to 28.2] | 11.4 [3.8 to 24.6] | 5.3 [1.5 to 13.1]
  Redness: Severe: number analyzed (Participants) | 47 | 85 | 42 | 73
  Redness: Severe | 0.0 [0.0 to 7.5] | 10.6 [5.0 to 19.2] | 2.4 [0.1 to 12.6] | 1.4 [0.0 to 7.4]
  Swelling: Any: number analyzed (Participants) | 53 | 104 | 49 | 84
  Swelling: Any | 24.5 [13.8 to 38.3] | 35.6 [26.4 to 45.6] | 20.4 [10.2 to 34.3] | 22.6 [14.2 to 33.0]
  Swelling: Mild: number analyzed (Participants) | 52 | 91 | 48 | 84
  Swelling: Mild | 21.2 [11.1 to 34.7] | 20.9 [13.1 to 30.7] | 18.8 [8.9 to 32.6] | 21.4 [13.2 to 31.7]
  Swelling: Moderate: number analyzed (Participants) | 49 | 95 | 43 | 73
  Swelling: Moderate | 10.2 [3.4 to 22.2] | 24.2 [16.0 to 34.1] | 7.0 [1.5 to 19.1] | 4.1 [0.9 to 11.5]
  Swelling: Severe: number analyzed (Participants) | 47 | 82 | 42 | 73
  Swelling: Severe | 0.0 [0.0 to 7.5] | 7.3 [2.7 to 15.2] | 2.4 [0.1 to 12.6] | 1.4 [0.0 to 7.4]
  Pain: Any: number analyzed (Participants) | 79 | 164 | 87 | 173
  Pain: Any | 78.5 [67.8 to 86.9] | 84.8 [78.3 to 89.9] | 83.9 [74.5 to 90.9] | 93.1 [88.2 to 96.4]
  Pain: Mild: number analyzed (Participants) | 76 | 156 | 83 | 165
  Pain: Mild | 76.3 [65.2 to 85.3] | 80.1 [73.0 to 86.1] | 81.9 [72.0 to 89.5] | 90.9 [85.4 to 94.8]
  Pain: Moderate: number analyzed (Participants) | 53 | 111 | 59 | 112
  Pain: Moderate | 24.5 [13.8 to 38.3] | 51.4 [41.7 to 61.0] | 44.1 [31.2 to 57.6] | 53.6 [43.9 to 63.0]
  Pain: Severe: number analyzed (Participants) | 48 | 86 | 44 | 75
  Pain: Severe | 2.1 [0.1 to 11.1] | 11.6 [5.7 to 20.3] | 9.1 [2.5 to 21.7] | 5.3 [1.5 to 13.1]
  Limitation of arm movement: Any: number analyzed (Participants) | 54 | 112 | 57 | 109
  Limitation of arm movement: Any | 27.8 [16.5 to 41.6] | 48.2 [38.7 to 57.9] | 42.1 [29.1 to 55.9] | 51.4 [41.6 to 61.1]
  Limitation of arm movement: Mild: number analyzed (Participants) | 54 | 110 | 57 | 106
  Limitation of arm movement: Mild | 24.1 [13.5 to 37.6] | 46.4 [36.8 to 56.1] | 40.4 [27.6 to 54.2] | 48.1 [38.3 to 58.0]
  Limitation of arm movement:Moderate: number analyzed (Participants) | 47 | 81 | 43 | 77
  Limitation of arm movement:Moderate | 4.3 [0.5 to 14.5] | 3.7 [0.8 to 10.4] | 7.0 [1.5 to 19.1] | 9.1 [3.7 to 17.8]
  Limitation of arm movement: Severe: number analyzed (Participants) | 47 | 84 | 41 | 77
  Limitation of arm movement: Severe | 2.1 [0.1 to 11.3] | 9.5 [4.2 to 17.9] | 4.9 [0.6 to 16.5] | 5.2 [1.4 to 12.8]

2. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 2 (Year 3 to 4) in Cohort 1 and Cohort 2
Description: Systemic events reported using an electronic diary. Systemic events are any fever >=38 degrees C, fatigue, headache, chills, rash, vomiting, decreased appetite, new generalized muscle pain, aggravated generalized muscle pain , new generalized joint pain), and aggravated generalized joint pain.
Time Frame: Within 14 days after vaccination 2
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants with known values for any systemic events. 'n'=number of participants with known values for specified systemic events for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 23vPS/23vPS, Cohort 1: Participants 60-64 years of age who received 23vPS at vaccination 1, received a 0.5 mL single dose intramuscularly of open-label 23vPS (Vaccination 2) at Year 3 to 4.
- 13vPnC/23vPS, Cohort 1: Participants 60-64 years of age who received 13vPnC at vaccination 1, received a 0.5 mL single dose of open-label 23vPS (Vaccination 2) at Year 3 to 4.
Arm/Group | 13vPnC/13vPnC, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Number analyzed (Participants) | 80 | 162 | 83 | 167
Percentage of participants
  Fever >=38 degrees C: number analyzed (Participants) | 48 | 79 | 43 | 75
  Fever >=38 degrees C | 2.1 [0.1 to 11.1] | 2.5 [0.3 to 8.8] | 4.7 [0.6 to 15.8] | 2.7 [0.3 to 9.3]
  Fever >= 38 to <38.5 degrees C: number analyzed (Participants) | 47 | 79 | 42 | 75
  Fever >= 38 to <38.5 degrees C | 0.0 [0.0 to 7.5] | 2.5 [0.3 to 8.8] | 2.4 [0.1 to 12.6] | 2.7 [0.3 to 9.3]
  Fever >=38.5 to <39 degrees C: number analyzed (Participants) | 48 | 78 | 42 | 73
  Fever >=38.5 to <39 degrees C | 2.1 [0.1 to 11.1] | 0.0 [0.0 to 4.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 4.9]
  Fever >=39 to =<40 degrees C: number analyzed (Participants) | 47 | 78 | 41 | 73
  Fever >=39 to =<40 degrees C | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 4.6] | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 4.9]
  Fever >40 degrees C: number analyzed (Participants) | 47 | 78 | 41 | 73
  Fever >40 degrees C | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 4.6] | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 4.9]
  Fatigue: number analyzed (Participants) | 69 | 125 | 68 | 125
  Fatigue | 50.7 [38.4 to 63.03] | 57.6 [48.4 to 66.4] | 63.2 [50.7 to 74.6] | 60.8 [51.7 to 69.4]
  Headache: number analyzed (Participants) | 60 | 118 | 64 | 123
  Headache | 38.3 [26.1 to 51.8] | 54.2 [44.8 to 63.4] | 50.0 [37.2 to 62.8] | 61.8 [52.6 to 70.4]
  Chills: number analyzed (Participants) | 52 | 99 | 56 | 93
  Chills | 23.1 [12.5 to 36.8] | 34.3 [25.1 to 44.6] | 33.9 [21.8 to 47.8] | 25.8 [17.3 to 35.9]
  Rash: number analyzed (Participants) | 51 | 95 | 49 | 81
  Rash | 23.5 [12.8 to 37.5] | 32.6 [23.4 to 43.0] | 18.4 [8.8 to 32.0] | 13.6 [7.0 to 23.0]
  Vomiting: number analyzed (Participants) | 48 | 79 | 43 | 76
  Vomiting | 8.3 [2.3 to 20.0] | 1.3 [0.0 to 6.9] | 4.7 [0.6 to 15.8] | 3.9 [0.8 to 11.1]
  Decreased appetite: number analyzed (Participants) | 52 | 93 | 54 | 89
  Decreased appetite | 21.2 [11.1 to 34.7] | 23.7 [15.5 to 33.6] | 31.5 [19.5 to 45.6] | 24.7 [16.2 to 35.0]
  New generalized muscle pain: number analyzed (Participants) | 60 | 136 | 66 | 128
  New generalized muscle pain | 55.0 [41.6 to 67.9] | 67.6 [59.1 to 75.4] | 65.2 [52.4 to 76.5] | 69.5 [60.8 to 77.4]
  Aggravated generalized muscle pain: number analyzed (Participants) | 51 | 101 | 58 | 95
  Aggravated generalized muscle pain | 27.5 [15.9 to 41.7] | 39.6 [30.0 to 49.8] | 41.4 [28.6 to 55.1] | 34.7 [25.3 to 45.2]
  New generalized joint pain: number analyzed (Participants) | 53 | 91 | 53 | 93
  New generalized joint pain | 18.9 [9.4 to 32.0] | 23.1 [14.9 to 33.1] | 24.5 [13.8 to 38.3] | 33.3 [23.9 to 43.9]
  Aggravated generalized joint pain: number analyzed (Participants) | 51 | 91 | 49 | 88
  Aggravated generalized joint pain | 13.7 [5.7 to 26.3] | 17.6 [10.4 to 27.0] | 22.4 [11.8 to 36.6] | 25.0 [16.4 to 35.4]

3. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Vaccination 1
Description: Serotype-specific OPA GMTs for the 13 pneumococcal common serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using microcolony OPA (mcOPA) assay. CIs for GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: One month after vaccination 1
Population: Evaluable immunogenicity population:eligible participants, received vaccination to which randomized, blood drawn within required timeframes, at least 1 valid, determinate assay result for proposed analysis, received no prohibited vaccines, no major protocol violations. n= number of participants with determinate OPA antibody titer to given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 23vPS, Cohort 1: Participants 60-64 years of age received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose intramuscularly (Vaccination 1).
- 13vPnC, Cohort 2: Participants 50-59 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly at (Vaccination 1).
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3
Number analyzed (Participants) | 411 | 407 | 388 | 874
titer
  1: number analyzed (Participants) | 404 | 402 | 382 | 866
  1 | 146 [124.0 to 172.9] | 104 [87.7 to 124.4] | 200 [170.3 to 236.0] | 353 [322.8 to 386.9]
  3: number analyzed (Participants) | 394 | 401 | 379 | 860
  3 | 93 [81.1 to 106.6] | 85 [74.2 to 98.3] | 91 [79.9 to 104.7] | 91 [84.2 to 98.4]
  4: number analyzed (Participants) | 359 | 367 | 350 | 849
  4 | 2062 [1693.6 to 2510.5] | 1295 [1045.9 to 1603.0] | 2833 [2412.1 to 3327.4] | 4747 [4370.2 to 5155.5]
  5: number analyzed (Participants) | 392 | 393 | 373 | 836
  5 | 199 [164.0 to 242.3] | 162 [133.6 to 197.5] | 269 [218.1 to 332.5] | 386 [342.6 to 435.8]
  6A: number analyzed (Participants) | 401 | 392 | 384 | 855
  6A | 2593 [2146.7 to 3131.1] | 213 [160.3 to 284.3] | 4328 [3658.1 to 5121.5] | 5746 [5240.7 to 6300.4]
  6B: number analyzed (Participants) | 371 | 371 | 361 | 865
  6B | 1984 [1604.0 to 2453.6] | 788 [615.9 to 1008.5] | 3212 [2728.6 to 3781.4] | 9813 [9097.8 to 10583.5]
  7F: number analyzed (Participants) | 394 | 396 | 378 | 859
  7F | 1120 [907.6 to 1382.9] | 405 [311.9 to 524.7] | 1520 [1274.5 to 1812.1] | 3249 [2994.8 to 3523.9]
  9V: number analyzed (Participants) | 367 | 368 | 364 | 844
  9V | 1164 [934.8 to 1448.3] | 407 [307.2 to 539.8] | 1726 [1428.5 to 2086.2] | 3339 [3037.4 to 3670.4]
  14: number analyzed (Participants) | 375 | 378 | 373 | 860
  14 | 612 [489.6 to 764.2] | 692 [553.3 to 866.2] | 957 [779.6 to 1174.5] | 2983 [2740.5 to 3246.6]
  18C: number analyzed (Participants) | 379 | 381 | 373 | 850
  18C | 1726 [1429.7 to 2082.9] | 925 [735.3 to 1162.9] | 1939 [1599.2 to 2350.2] | 3989 [3629.4 to 4383.8]
  19A: number analyzed (Participants) | 392 | 388 | 377 | 855
  19A | 682 [596.5 to 779.9] | 352 [297.0 to 416.1] | 956 [837.6 to 1090.7] | 1580 [1471.4 to 1696.3]
  19F: number analyzed (Participants) | 377 | 370 | 367 | 841
  19F | 517 [420.8 to 635.3] | 539 [442.1 to 658.2] | 599 [491.0 to 731.0] | 1533 [1397.3 to 1680.9]
  23F: number analyzed (Participants) | 375 | 375 | 368 | 851
  23F | 375 [297.2 to 472.6] | 72 [55.9 to 93.4] | 494 [386.8 to 630.7] | 1570 [1392.8 to 1770.2]
Statistical Analysis 1: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.10 to 1.78]
Statistical Analysis 2: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.1, 95% CI 2-sided [0.90 to 1.32]
Statistical Analysis 3: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.6, 95% CI 2-sided [1.19 to 2.13]
Statistical Analysis 4: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.2, 95% CI 2-sided [0.93 to 1.62]
Statistical Analysis 5: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 12.1, 95% CI 2-sided [8.63 to 17.08]
Statistical Analysis 6: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.5, 95% CI 2-sided [1.82 to 3.48]
Statistical Analysis 7: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.8, 95% CI 2-sided [1.98 to 3.87]
Statistical Analysis 8: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.9, 95% CI 2-sided [2.00 to 4.08]
Statistical Analysis 9: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.9, 95% CI 2-sided [0.64 to 1.21]
Statistical Analysis 10: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.9, 95% CI 2-sided [1.39 to 2.51]
Statistical Analysis 11: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.9, 95% CI 2-sided [1.56 to 2.41]
Statistical Analysis 12: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.0, 95% CI 2-sided [0.72 to 1.28]
Statistical Analysis 13: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 5.2, 95% CI 2-sided [3.67 to 7.33]
Statistical Analysis 14: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.08 to 1.73]
Statistical Analysis 15: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.0, 95% CI 2-sided [0.81 to 1.19]
Statistical Analysis 16: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.07 to 1.77]
Statistical Analysis 17: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI [1.01 to 1.80]
Statistical Analysis 18: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.7, 95% CI 2-sided [1.30 to 2.15]
Statistical Analysis 19: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.6, 95% CI 2-sided [1.24 to 2.12]
Statistical Analysis 20: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.03 to 1.79]
Statistical Analysis 21: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.5, 95% CI [1.11 to 1.98]
Statistical Analysis 22: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.6, 95% CI 2-sided [1.16 to 2.12]
Statistical Analysis 23: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.1, 95% CI 2-sided [0.86 to 1.47]
Statistical Analysis 24: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.16 to 1.69]
Statistical Analysis 25: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.2, 95% CI 2-sided [0.87 to 1.54]
Statistical Analysis 26: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.3, 95% CI 2-sided [0.94 to 1.84]
Statistical Analysis 27: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.4, 95% CI 2-sided [2.03 to 2.87]
Statistical Analysis 28: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.0, 95% CI 2-sided [0.84 to 1.13]
Statistical Analysis 29: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.3, 95% CI 2-sided [1.92 to 2.76]
Statistical Analysis 30: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.9, 95% CI 2-sided [1.55 to 2.42]
Statistical Analysis 31: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.2, 95% CI 2-sided [1.84 to 2.67]
Statistical Analysis 32: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.9, 95% CI 2-sided [4.13 to 5.93]
Statistical Analysis 33: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.9, 95% CI 2-sided [2.41 to 3.49]
Statistical Analysis 34: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.9, 95% CI 2-sided [2.34 to 3.52]
Statistical Analysis 35: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.9, 95% CI 2-sided [4.01 to 5.93]
Statistical Analysis 36: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.3, 95% CI 2-sided [1.91 to 2.79]
Statistical Analysis 37: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.3, 95% CI 2-sided [2.02 to 2.66]
Statistical Analysis 38: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.0, 95% CI 2-sided [2.44 to 3.60]
Statistical Analysis 39: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures in 13vPnC participants between Cohort 1 and Cohort 3; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.2, 95% CI 2-sided [3.31 to 5.31]

4. Primary Outcome: Percentage of Participants Achieving At Least a 4-fold Rise in OPA Titer for Serotype 6A 1 Month After Vaccination 1 in Cohort 1
Description: For serotype 6A the percentage of participants achieving at least a 4-fold rise on the serotype-specific antibody titer from pre-vaccination to 1 month post-vaccination was computed along with exact, 2-sided 95% confidence interval for the proportion.
Time Frame: One month after vaccination 1
Population: Evaluable immunogenicity population; N (number of participants analyzed) signifies participants with determinate OPA antibody titer to serotype 6A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1
Number analyzed (Participants) | 374 | 377
percentage of participants | 88.5 [84.8 to 91.6] | 49.3 [44.2 to 54.5]
Statistical Analysis 1: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; Difference in Percentage = 39.2, 95% CI 2-sided [33.0 to 45.1]

5. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Vaccination for 12 Common Serotypes in 13vPnC/23vPS Group Relative to 23vPS Group and 23vPS/23vPS Group
Description: Serotype-specific OPA GMTs for the 12 pneumococcal common serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using mcOPA assay. CIs for GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: One month after vaccination 1 and One month after vaccination 2/Year 3 to 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC/23vPS, Cohort 1 | 23vPS, Cohort 1 | 23vPs/23vPS, Cohort 1
Number analyzed (Participants) | 108 | 407 | 189
titers
  1: number analyzed (Participants) | 105 | 184 | 186
  1 | 398 [306.2 to 516.3] | 116 [89.4 to 149.6] | 95 [74.8 to 121.1]
  3: number analyzed (Participants) | 107 | 184 | 181
  3 | 164 [129.0 to 207.5] | 105 [85.3 to 128.7] | 53 [42.8 to 64.4]
  4: number analyzed (Participants) | 107 | 174 | 174
  4 | 1875 [1488.8 to 2360.7] | 1420 [1066.2 to 1890.5] | 733 [555.1 to 968.2]
  5: number analyzed (Participants) | 106 | 181 | 180
  5 | 476 [356.2 to 636.1] | 149 [111.1 to 201.2] | 74 [54.2 to 100.3]
  6B: number analyzed (Participants) | 104 | 174 | 181
  6B | 2670 [2012.9 to 3540.6] | 1088 [774.7 to 1528.1] | 916 [670.0 to 1252.4]
  7F: number analyzed (Participants) | 105 | 181 | 182
  7F | 1895 [1471.0 to 2441.1] | 403 [276.3 to 588.9] | 497 [361.8 to 682.0]
  9V: number analyzed (Participants) | 107 | 167 | 177
  9V | 1089 [699.2 to 1695.0] | 654 [452.5 to 944.9] | 187 [125.0 to 280.3]
  14: number analyzed (Participants) | 105 | 173 | 180
  14 | 1268 [951.8 to 1690.0] | 824 [612.9 to 1107.8] | 661 [515.6 to 848.6]
  18C: number analyzed (Participants) | 103 | 174 | 180
  18C | 2489 [1941.1 to 3192.7] | 1135 [815.7 to 1578.6] | 802 [597.5 to 1076.8]
  19A: number analyzed (Participants) | 106 | 182 | 184
  19A | 966 [763.2 to 1223.6] | 377 [296.1 to 479.6] | 364 [290.0 to 458.0]
  19F: number analyzed (Participants) | 99 | 170 | 176
  19F | 1653 [1302.2 to 2099.5] | 621 [468.6 to 821.7] | 374 [286.1 to 488.2]
  23F: number analyzed (Participants) | 105 | 173 | 181
  23F | 299 [203.9 to 437.5] | 86 [58.8 to 124.5] | 54 [38.4 to 77.0]
Statistical Analysis 1: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.4, 95% CI 2-sided [2.32 to 5.09]
Statistical Analysis 2: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.6, 95% CI 2-sided [1.13 to 2.16]
Statistical Analysis 3: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.3, 95% CI 2-sided [0.88 to 1.98]
Statistical Analysis 4: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.2, 95% CI 2-sided [2.04 to 4.97]
Statistical Analysis 5: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.5, 95% CI 2-sided [1.50 to 4.00]
Statistical Analysis 6: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.7, 95% CI 2-sided [2.76 to 7.99]
Statistical Analysis 7: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.7, 95% CI 2-sided [0.93 to 2.97]
Statistical Analysis 8: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.5, 95% CI 2-sided [0.99 to 2.39]
Statistical Analysis 9: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.2, 95% CI 2-sided [1.37 to 3.50]
Statistical Analysis 10: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.6, 95% CI 2-sided [1.78 to 3.68]
Statistical Analysis 11: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.7, 95% CI 2-sided [1.77 to 4.01]
Statistical Analysis 12: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.5, 95% CI 2-sided [1.99 to 6.13]
Statistical Analysis 13: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.2, 95% CI 2-sided [2.87 to 6.08]
Statistical Analysis 14: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.1, 95% CI 2-sided [2.26 to 4.30]
Statistical Analysis 15: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT ratio = 2.6, 95% CI 2-sided [1.72 to 3.80]
Statistical Analysis 16: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 6.5, 95% CI 2-sided [4.09 to 10.19]
Statistical Analysis 17: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.9, 95% CI 2-sided [1.83 to 4.63]
Statistical Analysis 18: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.8, 95% CI 2-sided [2.41 to 6.03]
Statistical Analysis 19: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 5.8, 95% CI 2-sided [3.13 to 10.82]
Statistical Analysis 20: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.9, 95% CI 2-sided [1.30 to 2.84]
Statistical Analysis 21: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 3.1, 95% CI 2-sided [2.02 to 4.78]
Statistical Analysis 22: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.7, 95% CI 2-sided [1.87 to 3.76]
Statistical Analysis 23: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 4.4, 95% CI 2-sided [2.97 to 6.58]
Statistical Analysis 24: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 5.5, 95% CI 2-sided [3.20 to 9.41]

6. Secondary Outcome: Percentage of Participants Achieving OPA Titers With at Least Lower Limit of Quantification (LLOQ) 1 Month After Vaccination 1
Description: Percentage of participants achieving OPA GMTs with at least LLOQ for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) determined in blood samples of all participants using mcOPA assay. Exact 2-sided CI based on observed proportion of participants. LLOQ for each serotype: 1=1:18, 3=1:12, 4=1:21, 5=1:29, 6A=1:37, 6B=1:43, 7F=1:210, 9V=1:345, 14=1:35, 18C=1:31, 19A=1:18, 19F=1:48, 23F=1:13.
Time Frame: One month after vaccination 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3
Number analyzed (Participants) | 411 | 407 | 388 | 874
Percentage of participants
  1: number analyzed (Participants) | 404 | 402 | 382 | 866
  1 | 90.3 [87.0 to 93.0] | 83.8 [79.9 to 87.3] | 94.0 [91.1 to 96.1] | 97.6 [96.3 to 98.5]
  3: number analyzed (Participants) | 394 | 401 | 379 | 860
  3 | 92.1 [89.0 to 94.6] | 88.3 [84.7 to 91.3] | 92.3 [89.2 to 94.8] | 94.8 [93.1 to 96.2]
  4: number analyzed (Participants) | 359 | 367 | 350 | 849
  4 | 95.0 [92.2 to 97.0] | 91.6 [88.2 to 94.2] | 97.4 [95.2 to 98.8] | 99.2 [98.3 to 99.7]
  5: number analyzed (Participants) | 392 | 393 | 373 | 836
  5 | 87.0 [83.3 to 90.2] | 84.7 [80.8 to 88.1] | 86.1 [82.1 to 89.4] | 92.1 [90.1 to 93.8]
  6A: number analyzed (Participants) | 401 | 392 | 384 | 855
  6A | 95.8 [93.3 to 97.5] | 69.1 [64.3 to 73.7] | 97.9 [95.9 to 99.1] | 99.4 [98.6 to 99.8]
  6B: number analyzed (Participants) | 371 | 371 | 361 | 865
  6B | 93.5 [90.5 to 95.8] | 86.0 [82.0 to 89.4] | 97.5 [95.3 to 98.9] | 99.9 [99.4 to 100.0]
  7F: number analyzed (Participants) | 394 | 396 | 378 | 859
  7F | 90.4 [87.0 to 93.1] | 78.0 [73.6 to 82.0] | 94.7 [91.9 to 96.7] | 98.6 [97.6 to 99.3]
  9V: number analyzed (Participants) | 367 | 368 | 364 | 844
  9V | 89.9 [86.4 to 92.8] | 75.8 [71.1 to 80.1] | 93.7 [90.7 to 96.0] | 97.7 [96.5 to 98.6]
  14: number analyzed (Participants) | 375 | 378 | 373 | 860
  14 | 87.7 [84.0 to 90.9] | 88.6 [85.0 to 91.6] | 92.0 [88.7 to 94.5] | 99.0 [98.0 to 99.5]
  18C: number analyzed (Participants) | 379 | 381 | 373 | 850
  18C | 95.5 [92.9 to 97.4] | 89.0 [85.4 to 91.9] | 94.9 [92.2 to 96.9] | 98.6 [97.5 to 99.3]
  19A: number analyzed (Participants) | 392 | 388 | 377 | 855
  19A | 98.5 [96.7 to 99.4] | 94.3 [91.5 to 96.4] | 98.4 [96.6 to 99.4] | 99.9 [99.4 to 100.0]
  19F: number analyzed (Participants) | 377 | 370 | 367 | 841
  19F | 89.7 [86.1 to 92.5] | 90.8 [87.4 to 93.6] | 91.6 [88.2 to 94.2] | 98.1 [96.9 to 98.9]
  23F: number analyzed (Participants) | 375 | 375 | 368 | 851
  23F | 84.5 [80.5 to 88.0] | 61.3 [56.2 to 66.3] | 85.1 [81.0 to 88.5] | 95.1 [93.4 to 96.4]
Statistical Analysis 1: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 1: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 6.5, 95% CI 2-sided [1.9 to 11.2]
Statistical Analysis 2: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 3: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.9, 95% CI 2-sided [-0.3 to 8.1]
Statistical Analysis 3: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 4: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.4, 95% CI 2-sided [-0.2 to 7.2]
Statistical Analysis 4: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 5: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 2.3, 95% CI 2-sided [-2.6 to 7.2]
Statistical Analysis 5: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 6A: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 26.6, 95% CI 2-sided [21.7 to 31.7]
Statistical Analysis 6: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 6B: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 7.5, 95% CI 2-sided [3.2 to 12.0]
Statistical Analysis 7: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 7F: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 12.3, 95% CI 2-sided [7.3 to 17.4]
Statistical Analysis 8: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 9V: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 14.1, 95% CI 2-sided [8.7 to 19.5]
Statistical Analysis 9: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 14: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = -0.9, 95% CI 2-sided [-5.6 to 3.8]
Statistical Analysis 10: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 18C: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 6.5, 95% CI 2-sided [2.6 to 10.5]
Statistical Analysis 11: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 19A: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 4.1, 95% CI 2-sided [1.2 to 7.1]
Statistical Analysis 12: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; Difference in Percentage = -1.2, 95% CI 2-sided [-5.5 to 3.2]
Statistical Analysis 13: Comparison: 13vPnC, Cohort 1 vs 23vPS, Cohort 1; Serotype 23F: Difference (13vPnC - 23vPS) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 23.2, 95% CI 2-sided [17.0 to 29.3]
Statistical Analysis 14: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 1: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.6, 95% CI 2-sided [-0.2 to 7.5]
Statistical Analysis 15: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 3: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 0.2, 95% CI 2-sided [-3.6 to 4.1]
Statistical Analysis 16: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 4: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 2.4, 95% CI 2-sided [-0.4 to 5.5]
Statistical Analysis 17: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 5: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = -0.9, 95% CI 2-sided [-5.8 to 3.9]
Statistical Analysis 18: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 6A: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 2.2, 95% CI 2-sided [-0.4 to 4.8]
Statistical Analysis 19: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 6B: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 4.0, 95% CI 2-sided [0.8 to 7.2]
Statistical Analysis 20: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 7F: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 4.4, 95% CI 2-sided [0.6 to 8.2]
Statistical Analysis 21: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 9V: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.8, 95% CI 2-sided [-0.3 to 7.9]
Statistical Analysis 22: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 14: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Perecentage = 4.2, 95% CI 2-sided [-0.1 to 8.7]
Statistical Analysis 23: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 18C: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = -0.6, 95% CI 2-sided [-3.8 to 2.5]
Statistical Analysis 24: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 19A: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = -0.1, 95% CI 2-sided [-2.1 to 1.9]
Statistical Analysis 25: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 19F: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 1.9, 95% CI 2-sided [-2.4 to 6.2]
Statistical Analysis 26: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 2; Serotype 23F: Difference (cohort 2 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 0.5, 95% CI 2-sided [-4.7 to 5.7]
Statistical Analysis 27: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 1: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 7.2, 95% CI 2-sided [4.3 to 10.6]
Statistical Analysis 28: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 3: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 2.6, 95% CI 2-sided [-0.3 to 5.9]
Statistical Analysis 29: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 4: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 4.2, 95% CI 2-sided [2.1 to 6.9]
Statistical Analysis 30: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 5: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 5.1, 95% CI 2-sided [1.4 to 9.1]
Statistical Analysis 31: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 6A: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.7, 95% CI 2-sided [1.7 to 6.1]
Statistical Analysis 32: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 6B: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 6.4, 95% CI 2-sided [4.1 to 9.3]
Statistical Analysis 33: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 7F: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 8.2, 95% CI 2-sided [5.4 to 11.6]
Statistical Analysis 34: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 9V: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 7.8, 95% CI 2-sided [4.8 to 11.4]
Statistical Analysis 35: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 14: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 11.2, 95% CI 2-sided [8.0 to 14.9]
Statistical Analysis 36: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 18C: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 3.1, 95% CI 2-sided [0.9 to 5.7]
Statistical Analysis 37: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 19A: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 1.4, 95% CI 2-sided [0.3 to 3.1]
Statistical Analysis 38: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 19F: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 8.4, 95% CI 2-sided [5.4 to 12.0]
Statistical Analysis 39: Comparison: 13vPnC, Cohort 1 vs 13vPnC, Cohort 3; Serotype 23F: Difference (cohort 3 - cohort 1) in proportions, expressed as a percentage presented along with exact 2-sided 95%CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than -0.10; Difference in Percentage = 10.5, 95% CI 2-sided [6.8 to 14.7]

7. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) for the 13 Serotypes From Prevaccination 1 to 1 Month After Vaccination 2 in Cohort 1 and Cohort 2
Description: Geometric mean fold rises (GMFRs) for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from prevaccination to 1 month postvaccination were computed using the logarithmically transformed assay results. CI for the GMFRs are back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: Prevaccination 1 to 1 month after vaccination 2/Year 3 to 4
Population: Evaluable immunogenicity population; n= number of participants with valid and determinate assay results for the specified serotype at both sampling times.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | 13vPnC/13vPnC, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 23vPS/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Number analyzed (Participants) | 108 | 108 | 189 | 211
Fold Rise
  1: number analyzed (Participants) | 102 | 103 | 185 | 202
  1 | 72.6 [53.90 to 97.82] | 69.7 [51.85 to 93.79] | 15.6 [12.38 to 19.73] | 54.0 [43.92 to 66.50]
  3: number analyzed (Participants) | 98 | 100 | 176 | 198
  3 | 13.2 [9.98 to 17.33] | 21.2 [15.46 to 29.15] | 6.8 [5.49 to 8.54] | 11.5 [9.51 to 13.91]
  4: number analyzed (Participants) | 85 | 87 | 136 | 165
  4 | 68.0 [40.04 to 115.58] | 110.4 [66.47 to 183.22] | 43.8 [27.87 to 68.74] | 104.2 [70.96 to 152.94]
  5: number analyzed (Participants) | 101 | 103 | 177 | 201
  5 | 47.9 [33.51 to 68.52] | 83.2 [60.56 to 114.26] | 11.9 [8.94 to 15.71] | 52.8 [41.81 to 66.71]
  6A: number analyzed (Participants) | 93 | 99 | 166 | 189
  6A | 142.0 [84.10 to 239.68] | 116.2 [71.19 to 189.69] | 6.4 [4.25 to 9.53] | 139.7 [93.99 to 207.79]
  6B: number analyzed (Participants) | 89 | 89 | 157 | 181
  6B | 103.3 [57.72 to 184.69] | 63.6 [34.73 to 116.29] | 24.9 [15.98 to 38.77] | 132.7 [84.86 to 207.38]
  7F: number analyzed (Participants) | 97 | 100 | 173 | 193
  7F | 140.8 [91.49 to 216.59] | 293.9 [203.35 to 424.67] | 72.1 [50.27 to 103.53] | 218.0 [169.33 to 280.62]
  9V: number analyzed (Participants) | 85 | 93 | 147 | 172
  9V | 24.7 [12.86 to 47.32] | 40.1 [21.13 to 76.11] | 10.6 [6.52 to 17.13] | 49.9 [32.88 to 75.68]
  14: number analyzed (Participants) | 95 | 97 | 165 | 189
  14 | 20.6 [12.31 to 34.57] | 36.6 [22.02 to 60.97] | 19.9 [13.85 to 28.67] | 26.6 [18.43 to 38.52]
  18C: number analyzed (Participants) | 95 | 97 | 170 | 191
  18C | 67.9 [41.02 to 112.48] | 80.9 [48.89 to 133.79] | 27.5 [19.10 to 39.69] | 94.9 [67.89 to 132.54]
  19A: number analyzed (Participants) | 96 | 93 | 168 | 196
  19A | 37.6 [25.57 to 55.37] | 43.1 [29.21 to 63.51] | 15.4 [11.79 to 20.25] | 30.9 [23.56 to 40.43]
  19F: number analyzed (Participants) | 93 | 93 | 160 | 186
  19F | 54.1 [34.08 to 86.01] | 110.3 [71.30 to 170.65] | 25.1 [18.04 to 34.84] | 60.4 [43.40 to 84.06]
  23F: number analyzed (Participants) | 95 | 97 | 169 | 188
  23F | 115.7 [77.40 to 172.81] | 32.5 [21.38 to 49.40] | 6.4 [4.57 to 8.85] | 130.0 [94.64 to 178.44]

8. Secondary Outcome: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) for 12 Common Serotypes in 13vPnC/23vPS Group Relative to 23vPS and 23vPS/23vPS Groups in Cohort 1; and in 13vPnC/13vPnC Group in Cohort 2, 1 Month After Vaccination
Description: Antibody geometric mean concentration (GMC) as measured by microgram/milliliter (mcg/mL) for 12 common pneumococcal serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: One month after vaccination 1 and One month after vaccination 2/Year 3 to 4
Population: Evaluable immunogenicity population; n= number of participants with a determinate IgG concentration to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- 13vPnC/13vPnC, Cohort 2: Participants 50-59 years of age who received 13vPnC at vaccination 1, received a 0.5 mL single dose intramuscularly of open-label 13vPnC (Vaccination 2) at Year 3 to 4.
Arm/Group | 13vPnC/23vPS, Cohort 1 | 23vPS, Cohort 1 | 23vPs/23vPS, Cohort 1 | 13vPnC/13vPnC, Cohort 2
Number analyzed (Participants) | 108 | 407 | 189 | 211
mcg/mL
  1: number analyzed (Participants) | 99 | 48 | 98 | 98
  1 | 9.53 [7.53 to 12.07] | 4.13 [2.86 to 5.96] | 4.36 [3.33 to 5.72] | 6.92 [5.31 to 9.03]
  3: number analyzed (Participants) | 99 | 46 | 98 | 98
  3 | 2.58 [2.14 to 3.11] | 1.88 [1.29 to 2.74] | 1.81 [1.44 to 2.29] | 1.33 [1.07 to 1.64]
  4: number analyzed (Participants) | 99 | 48 | 98 | 93
  4 | 3.68 [2.86 to 4.74] | 1.59 [1.06 to 2.37] | 1.49 [1.14 to 1.95] | 4.89 [3.83 to 6.25]
  5: number analyzed (Participants) | 99 | 47 | 98 | 97
  5 | 11.52 [9.09 to 14.61] | 8.23 [5.81 to 11.67] | 5.78 [4.66 to 7.16] | 7.23 [5.67 to 9.22]
  6B: number analyzed (Participants) | 98 | 47 | 98 | 97
  6B | 11.50 [9.21 to 14.37] | 7.81 [5.74 to 10.61] | 5.65 [4.58 to 6.97] | 19.07 [14.59 to 24.92]
  7F: number analyzed (Participants) | 98 | 47 | 97 | 95
  7F | 8.52 [6.83 to 10.62] | 8.24 [5.38 to 12.60] | 4.61 [3.57 to 5.95] | 6.26 [5.19 to 7.54]
  9V: number analyzed (Participants) | 99 | 47 | 97 | 97
  9V | 7.39 [5.99 to 9.10] | 5.50 [4.15 to 7.30] | 3.78 [3.07 to 4.65] | 4.97 [4.08 to 6.05]
  14: number analyzed (Participants) | 97 | 47 | 98 | 97
  14 | 16.07 [12.31 to 20.98] | 12.05 [7.26 to 19.99] | 8.22 [6.11 to 11.05] | 14.66 [11.97 to 17.96]
  18C: number analyzed (Participants) | 98 | 48 | 98 | 98
  18C | 8.56 [6.77 to 10.84] | 8.21 [5.64 to 11.96] | 6.30 [4.70 to 8.45] | 7.17 [5.68 to 9.03]
  19A: number analyzed (Participants) | 98 | 48 | 98 | 98
  19A | 14.63 [11.87 to 18.04] | 12.70 [9.29 to 17.37] | 9.88 [7.80 to 12.52] | 16.33 [13.31 to 20.04]
  19F: number analyzed (Participants) | 98 | 46 | 97 | 96
  19F | 11.51 [8.64 to 15.34] | 6.42 [4.11 to 10.01] | 3.44 [2.50 to 4.73] | 12.89 [9.75 to 17.06]
  23F: number analyzed (Participants) | 98 | 48 | 97 | 96
  23F | 7.11 [5.50 to 9.19] | 4.89 [3.52 to 6.81] | 3.56 [2.81 to 4.52] | 17.20 [13.28 to 22.29]
Statistical Analysis 1: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 1: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.31, 95% CI 2-sided [1.52 to 3.51]
Statistical Analysis 2: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 3: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.37, 95% CI 2-sided [0.95 to 1.99]
Statistical Analysis 3: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 4: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.32, 95% CI 2-sided [1.47 to 3.64]
Statistical Analysis 4: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 5: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.40, 95% CI 2-sided [0.92 to 2.12]
Statistical Analysis 5: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 6B: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.47, 95% CI 2-sided [1.01 to 2.16]
Statistical Analysis 6: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 7F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.03, 95% CI 2-sided [0.67 to 1.59]
Statistical Analysis 7: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 9V: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.34, 95% CI 2-sided [0.94 to 1.92]
Statistical Analysis 8: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 14: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.33, 95% CI 2-sided [0.80 to 2.23]
Statistical Analysis 9: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 18C: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.04, 95% CI 2-sided [0.68 to 1.59]
Statistical Analysis 10: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 19A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.15, 95% CI 2-sided [0.80 to 1.66]
Statistical Analysis 11: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 19F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.79, 95% CI [1.07 to 3.00]
Statistical Analysis 12: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPS, Cohort 1; Serotype 23F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.45, 95% CI 2-sided [0.95 to 2.24]
Statistical Analysis 13: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 1: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.18, 95% CI 2-sided [1.53 to 3.12]
Statistical Analysis 14: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 3: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.42, 95% CI 2-sided [1.06 to 1.91]
Statistical Analysis 15: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 4: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.47, 95% CI 2-sided [1.71 to 3.55]
Statistical Analysis 16: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 5: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.99, 95% CI 2-sided [1.45 to 2.74]
Statistical Analysis 17: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 6B: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.04, 95% CI 2-sided [1.50 to 2.76]
Statistical Analysis 18: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 7F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.85, 95% CI 2-sided [1.32 to 2.58]
Statistical Analysis 19: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 9V: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.96, 95% CI 2-sided [1.46 to 2.62]
Statistical Analysis 20: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 14: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.96, 95% CI 2-sided [1.32 to 2.91]
Statistical Analysis 21: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 18C: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.36, 95% CI 2-sided [0.94 to 1.97]
Statistical Analysis 22: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 19A: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 1.48, 95% CI 2-sided [1.08 to 2.03]
Statistical Analysis 23: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 19F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 3.35, 95% CI 2-sided [2.19 to 5.12]
Statistical Analysis 24: Comparison: 13vPnC/23vPS, Cohort 1 vs 23vPs/23vPS, Cohort 1; Serotype 23F: CI for the GMC ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC/23vPS - 23vPS/23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMC Ratio = 2.00, 95% CI 2-sided [1.41 to 2.83]

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 1
Description: Local reactions reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 centimeters [cm]; Moderate (5.1 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating); Limitation of arm movement scaled as Any (limitation [lim] present); Mild (some limitation); Moderate (unable to move arm above head; able to move arm above shoulder); Severe (unable to move arm above shoulder).
Time Frame: Within 14 days after vaccination 1
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed )=participants with known values for any local reaction. 'n'=number of participants with known values for specified local reaction for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 23vPS, Cohort 1: Participants 60-64 years of age received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose (Vaccination 1).
- 13vPnC, Cohort 2: Participants 50-59 years of age received 13vPnC administered as a 0.5 mL single dose at (Vaccination 1).
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3
Number analyzed (Participants) | 337 | 307 | 327 | 801
Percentage of participants
  Redness: Any: number analyzed (Participants) | 193 | 190 | 152 | 266
  Redness: Any | 20.2 [14.8 to 26.6] | 14.2 [9.6 to 20.0] | 15.8 [10.4 to 22.6] | 30.5 [25.0 to 36.4]
  Redness: Mild: number analyzed (Participants) | 189 | 187 | 151 | 258
  Redness: Mild | 15.9 [11.0 to 21.9] | 11.2 [7.1 to 16.7] | 15.2 [9.9 to 22.0] | 26.4 [21.1 to 32.2]
  Redness: Moderate: number analyzed (Participants) | 185 | 182 | 140 | 227
  Redness: Moderate | 8.6 [5.0 to 13.7] | 4.9 [2.3 to 9.2] | 5.0 [2.0 to 10.0] | 11.9 [8.0 to 16.8]
  Redness: Severe: number analyzed (Participants) | 178 | 179 | 137 | 211
  Redness: Severe | 1.7 [0.3 to 4.8] | 0.0 [0.0 to 0.2] | 0.7 [0.0 to 4.0] | 2.8 [1.1 to 6.1]
  Swelling: Any: number analyzed (Participants) | 197 | 191 | 161 | 302
  Swelling: Any | 19.3 [14.0 to 25.5] | 13.1 [8.7 to 18.7] | 21.7 [15.6 to 28.9] | 39.4 [33.9 to 45.2]
  Swelling: Mild: number analyzed (Participants) | 192 | 189 | 160 | 293
  Swelling: Mild | 15.6 [10.8 to 21.5] | 10.1 [6.2 to 15.3] | 20.6 [14.6 to 27.7] | 37.2 [31.7 to 43.0]
  Swelling: Moderate: number analyzed (Participants) | 184 | 181 | 138 | 238
  Swelling: Moderate | 8.2 [4.6 to 13.1] | 4.4 [1.9 to 8.5] | 4.3 [1.6 to 9.2] | 15.1 [10.8 to 20.3]
  Swelling: Severe: number analyzed (Participants) | 178 | 180 | 136 | 209
  Swelling: Severe | 0.6 [0.0 to 3.1] | 1.1 [0.1 to 4.0] | 0.0 [0.0 to 2.7] | 1.4 [0.3 to 4.1]
  Pain: Any: number analyzed (Participants) | 331 | 301 | 322 | 787
  Pain: Any | 80.1 [75.3 to 84.2] | 73.4 [68.1 to 78.3] | 88.8 [84.9 to 92.0] | 96.7 [95.2 to 97.8]
  Pain: Mild: number analyzed (Participants) | 323 | 290 | 306 | 721
  Pain: Mild | 78.6 [73.8 to 83.0] | 68.6 [62.9 to 73.9] | 85.9 [81.5 to 89.6] | 93.2 [91.1 to 94.4]
  Pain: Moderate: number analyzed (Participants) | 206 | 210 | 190 | 467
  Pain: Moderate | 23.3 [17.7 to 29.7] | 30.0 [23.9 to 36.7] | 39.5 [32.5 to 46.8] | 77.1 [73.0 to 80.8]
  Pain: Severe: number analyzed (Participants) | 178 | 187 | 139 | 238
  Pain: Severe | 1.7 [0.3 to 4.8] | 8.6 [5.0 to 13.5] | 3.6 [1.2 to 8.2] | 16.0 [11.6 to 21.3]
  Lim of arm movement:Any: number analyzed (Participants) | 214 | 211 | 194 | 499
  Lim of arm movement:Any | 28.5 [22.6 to 35.1] | 30.8 [24.6 to 37.5] | 40.7 [33.7 to 48.0] | 75.2 [71.1 to 78.9]
  Lim of arm movement:Mild: number analyzed (Participants) | 212 | 208 | 189 | 466
  Lim of arm movement:Mild | 26.9 [21.0 to 33.4] | 29.3 [23.2 to 36.0] | 38.6 [31.6 to 46.0] | 71.5 [67.1 to 75.5]
  Lim of arm movement:Moderate: number analyzed (Participants) | 179 | 182 | 140 | 238
  Lim of arm movement:Moderate | 2.2 [0.6 to 5.6] | 3.8 [1.6 to 7.8] | 2.9 [0.8 to 7.2] | 18.5 [13.8 to 24.0]
  Lim of arm movement:Severe: number analyzed (Participants) | 180 | 185 | 139 | 237
  Lim of arm movement:Severe | 1.7 [0.3 to 4.8] | 4.3 [1.9 to 8.3] | 2.9 [0.8 to 7.2] | 15.6 [11.2 to 20.9]

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 1
Description: Systemic events reported using an electronic diary. Systemic events are any fever greater than or equal to (>=) 38 degrees Celsius [C], fatigue, headache, chills, rash, vomiting, decreased appetite, new generalized (gen) muscle pain, aggravated generalized muscle pain , new generalized joint pain), and aggravated generalized joint pain. All reports of fever >40 degrees C in 13vPnC and 23vPS for Cohort 1 were confirmed as data entry errors.
Time Frame: Within 14 days after vaccination 1
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed )=participants with known values for any systemic events. 'n'=number of participants with known values for specified systemic events for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 13vPnC, Cohort 1: Participants 60-64 years of age received 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a 0.5 milliliter (mL) single dose intramuscularly (Vaccination 1 [Vax1]) at Year 0.
- 23vPS, Cohort 1: Participants 60-64 years of age received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose (Vaccination 1) at Year 0.
- 13vPnC, Cohort 2: Participants 50-59 years of age received 13vPnC administered as a 0.5 mL single dose at (Vaccination 1) Year 0.
Arm/Group | 13vPnC, Cohort 1 | 23vPS, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC, Cohort 3
Number analyzed (Participants) | 327 | 330 | 314 | 752
Percentage of participants
  Fever >=38 degrees C: number analyzed (Participants) | 181 | 185 | 137 | 221
  Fever >=38 degrees C | 7.7 [4.3 to 12.6] | 5.9 [3.0 to 10.4] | 1.5 [0.2 to 5.2] | 7.2 [4.2 to 11.5]
  Fever >=38 to <38.5 degrees C: number analyzed (Participants) | 179 | 180 | 137 | 214
  Fever >=38 to <38.5 degrees C | 3.9 [1.6 to 7.9] | 1.1 [0.1 to 4.0] | 1.5 [0.2 to 5.2] | 4.2 [1.9 to 7.8]
  Fever >=38.5 to <39 degrees C: number analyzed (Participants) | 178 | 179 | 136 | 211
  Fever >=38.5 to <39 degrees C | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.7] | 1.9 [0.5 to 4.8]
  Fever >=39 to =<40 degrees C: number analyzed (Participants) | 177 | 179 | 136 | 210
  Fever >=39 to =<40 degrees C | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.7] | 1.4 [0.3 to 4.1]
  Fever >40 degrees C: number analyzed (Participants) | 180 | 184 | 136 | 208
  Fever >40 degrees C | 4.4 [1.9 to 8.6] | 4.9 [2.3 to 9.1] | 0.0 [0.0 to 2.7] | 0.5 [0.0 to 2.6]
  Fatigue: number analyzed (Participants) | 277 | 273 | 248 | 554
  Fatigue | 63.2 [57.2 to 68.9] | 61.5 [55.5 to 67.3] | 63.3 [57.0 to 69.3] | 80.5 [77.0 to 83.7]
  Headache: number analyzed (Participants) | 252 | 259 | 246 | 527
  Headache | 54.0 [47.6 to 60.2] | 54.4 [48.2 to 60.6] | 65.9 [59.6 to 71.8] | 81.4 [77.8 to 84.6]
  Chills: number analyzed (Participants) | 204 | 199 | 158 | 286
  Chills | 23.5 [17.9 to 30.0] | 24.1 [18.4 to 30.7] | 19.6 [13.7 to 26.7] | 38.1 [32.5 to 44.0]
  Rash: number analyzed (Participants) | 194 | 192 | 148 | 249
  Rash | 16.5 [11.6 to 22.5] | 13.0 [8.6 to 18.6] | 14.2 [9.0 to 20.9] | 21.3 [16.4 to 26.9]
  Vomiting: number analyzed (Participants) | 180 | 186 | 144 | 240
  Vomiting | 3.9 [1.6 to 7.8] | 5.4 [2.6 to 9.7] | 6.9 [3.4 to 12.4] | 15.0 [10.7 to 20.2]
  Decreased appetite: number analyzed (Participants) | 202 | 207 | 166 | 363
  Decreased appetite | 21.3 [15.9 to 27.6] | 21.7 [16.3 to 28.0] | 25.3 [18.9 to 32.6] | 55.6 [50.4 to 60.8]
  New gen muscle pain: number analyzed (Participants) | 249 | 268 | 238 | 561
  New gen muscle pain | 56.2 [49.8 to 62.5] | 57.8 [51.7 to 63.8] | 61.8 [55.3 to 68.0] | 82.0 [78.6 to 85.1]
  Aggravated gen muscle pain: number analyzed (Participants) | 215 | 225 | 188 | 370
  Aggravated gen muscle pain | 32.6 [26.3 to 39.3] | 37.3 [31.0 to 44.0] | 39.9 [32.8 to 47.3] | 55.9 [50.7 to 61.1]
  New gen joint pain: number analyzed (Participants) | 197 | 216 | 165 | 307
  New gen joint pain | 24.4 [18.5 to 31.0] | 30.1 [24.1 to 36.7] | 31.5 [24.5 to 39.2] | 41.7 [36.1 to 47.4]
  Aggravated gen joint pain: number analyzed (Participants) | 205 | 206 | 168 | 269
  Aggravated gen joint pain | 24.9 [19.1 to 31.4] | 21.4 [16.0 to 27.6] | 25.6 [19.2 to 32.9] | 28.6 [23.3 to 34.4]

ADVERSE EVENTS:
Time Frame: Adverse events collected after vaccination and at the 6-month follow-up contact. Participants recorded pre-specified AEs in electronic diary: local reactions and systemic events from Day 1-Day 14 post vaccination.
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on the case report form at each visit (nonsystematic assessment).
Groups:
- 13vPnC, Cohort 1: Participants aged 60-64 years old received 13 valent pneumococcal conjugate (13vPnC) administered as a single dose 0.5 mL (Vaccination 1 [Vax1]), reported after vaccination.
- 13vPnC: 6 Month Follow-up After Vax 1, Cohort 1: Participants aged 60-64 years old received 13 valent pneumococcal conjugate (13vPnC) administered as a single dose 0.5 mL (Vaccination 1), reported at 6-month follow-up.
- 23vPS, Cohort 1: Participants aged 60-64 years old received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a single dose 0.5 mL (Vaccination 1), reported after vaccination 1.
- 23vPS: 6 Month Follow-up After Vax 1, Cohort 1: Participants aged 60-64 years old received 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a single dose 0.5 mL (Vaccination 1), reported at 6-month follow-up.
- 13vPnC, Cohort 2: Participants aged 50-59 years old received 13vPnC administered as a single dose 0.5 mL (Vaccination 1), reported after vaccination 1. Out of 404 participants vaccinated, 1 participant randomized and vaccinated in error without a consent form, and hence safety data is available for 403 participant.
- 13vPnC: 6 Month Follow-up After Vax 1, Cohort 2: Participants aged 50-59 years old received 13vPnC administered as a single dose 0.5 mL (Vaccination 1), reported at 6-month follow-up. Out of 404 participants vaccinated, 1 participant randomized and vaccinated in error without a consent form, and hence safety data is available for 403 participant.
- 13vPnC/13vPnC, Cohort 1: Participants aged 60-64 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 13vPnC at Year 3 to 4 (Vaccination 2), reported after vaccination 2.
- 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 1: Participants aged 60-64 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 13vPnC at Year 3 to 4 (Vaccination 2), reported at 6-month follow-up after vaccination 2.
- 13vPnC/23vPS, Cohort 1: Participants aged 60-64 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 23vPS at Year 3 to 4 (Vaccination 2), reported after vaccination 2.
- 13vPnC/23vPS: 6 Month Follow-up After Vax 2, Cohort 1: Participants aged 60-64 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 23vPS at Year 3 to 4 (Vaccination 2), reported at 6-month follow-up after vaccination 2.
- 23vPS/23vPS, Cohort 1: Participants aged 60-64 years old who received 23vPS at vaccination 1 received a 0.5 mL single dose of open-label 23vPS at Year 3 to 4 (Vaccination 2), reported after vaccination 2.
- 23vPS/23vPS: 6 Month Follow-up After Vax 2, Cohort 1: Participants aged 60-64 years old who received 23vPS at vaccination 1 received a 0.5 mL single dose of open-label 23vPS at Year 3 to 4 (Vaccination 2), reported at 6-month follow-up after vaccination 2.
- 13vPnC/13vPnC, Cohort 2: Participants aged 50-59 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 13vPnC at Year 3 to 4 (Vaccination 2), reported after vaccination 2.
- 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 2: Participants aged 50-59 years old who received 13vPnC at vaccination 1 received a 0.5 mL single dose of open-label 13vPnC at Year 3 to 4 (Vaccination 2), reported at 6-month follow-up after vaccination 2.
- 13vPnC, Cohort 3: Participants aged 18-49 years old received 13vPnC administered as a single dose 0.5 mL (Vaccination 1), reported after vaccination 1.
- 13vPnC: 6 Month Follow-up After Vax 1, Cohort 3: Participants aged 18-49 years old received 13vPnC administered as a single dose 0.5 mL (Vaccination 1), reported at 6-month follow-up.
Arm/Group | 13vPnC, Cohort 1 | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 1 | 23vPS, Cohort 1 | 23vPS: 6 Month Follow-up After Vax 1, Cohort 1 | 13vPnC, Cohort 2 | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 2 | 13vPnC/13vPnC, Cohort 1 | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 1 | 13vPnC/23vPS, Cohort 1 | 13vPnC/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 | 23vPS/23vPS, Cohort 1 | 23vPS/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 | 13vPnC/13vPnC, Cohort 2 | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 2 | 13vPnC, Cohort 3 | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 3
Serious Adverse Events (participants affected / at risk) | 1/417 | 12/417 | 2/414 | 10/414 | 2/403 | 5/403 | 1/108 | 2/108 | 1/108 | 1/108 | 0/189 | 3/189 | 0/214 | 0/214 | 2/899 | 2/899
Other Adverse Events (participants affected / at risk) | 277/417 | 0/417 | 271/414 | 5/414 | 293/403 | 2/403 | 66/108 | 1/108 | 73/108 | 4/108 | 143/189 | 13/189 | 164/214 | 4/214 | 779/899 | 1/899
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC, Cohort 1 (N=417) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 1 (N=417) | 23vPS, Cohort 1 (N=414) | 23vPS: 6 Month Follow-up After Vax 1, Cohort 1 (N=414) | 13vPnC, Cohort 2 (N=403) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 2 (N=403) | 13vPnC/13vPnC, Cohort 1 (N=108) | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 1 (N=108) | 13vPnC/23vPS, Cohort 1 (N=108) | 13vPnC/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 (N=108) | 23vPS/23vPS, Cohort 1 (N=189) | 23vPS/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 (N=189) | 13vPnC/13vPnC, Cohort 2 (N=214) | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 2 (N=214) | 13vPnC, Cohort 3 (N=899) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 3 (N=899)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 13vPnC, Cohort 1 (N=417) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 1 (N=417) | 23vPS, Cohort 1 (N=414) | 23vPS: 6 Month Follow-up After Vax 1, Cohort 1 (N=414) | 13vPnC, Cohort 2 (N=403) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 2 (N=403) | 13vPnC/13vPnC, Cohort 1 (N=108) | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 1 (N=108) | 13vPnC/23vPS, Cohort 1 (N=108) | 13vPnC/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 (N=108) | 23vPS/23vPS, Cohort 1 (N=189) | 23vPS/23vPS: 6 Month Follow-up After Vax 2, Cohort 1 (N=189) | 13vPnC/13vPnC, Cohort 2 (N=214) | 13vPnC/13vPnC: 6 Month Follow-up After Vax 2, Cohort 2 (N=214) | 13vPnC, Cohort 3 (N=899) | 13vPnC: 6 Month Follow-up After Vax 1, Cohort 3 (N=899)
Redness (Any) (Skin and subcutaneous tissue disorders) | 39/193 | 0/0 | 27/190 | 0/0 | 24/152 | 0/0 | 10/50 | 0/0 | 14/51 | 0/0 | 39/109 | 0/0 | 18/84 | 0/0 | 81/266 | 0
Redness (Mild) (Skin and subcutaneous tissue disorders) | 30/189 | 0/0 | 21/187 | 0/0 | 23/151 | 0/0 | 10/50 | 0/0 | 11/49 | 0/0 | 28/101 | 0/0 | 15/83 | 0/0 | 68/258 | 0
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 16/185 | 0/0 | 9/182 | 0/0 | 7/140 | 0/0 | 3/48 | 0/0 | 5/44 | 0/0 | 17/91 | 0/0 | 4/75 | 0/0 | 27/227 | 0
Redness (Severe) (Skin and subcutaneous tissue disorders) | 3/178 | 0/0 | 0/179 | 0/0 | 1/137 | 0/0 | 0/47 | 0/0 | 1/42 | 0/0 | 9/85 | 0/0 | 1/73 | 0/0 | 6/211 | 0
Swelling (Any) (Skin and subcutaneous tissue disorders) | 38/197 | 0/0 | 25/191 | 0/0 | 35/161 | 0/0 | 13/53 | 0/0 | 10/49 | 0/0 | 37/104 | 0/0 | 19/84 | 0/0 | 119/302 | 0
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 30/192 | 0/0 | 19/189 | 0/0 | 33/160 | 0/0 | 11/52 | 0/0 | 9/48 | 0/0 | 19/91 | 0/0 | 18/84 | 0/0 | 109/293 | 0
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 15/184 | 0/0 | 8/181 | 0/0 | 6/138 | 0/0 | 5/49 | 0/0 | 3/43 | 0/0 | 23/95 | 0/0 | 3/73 | 0/0 | 36/238 | 0
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/178 | 0/0 | 2/180 | 0/0 | 0/136 | 0/0 | 0/47 | 0/0 | 1/42 | 0/0 | 6/82 | 0/0 | 1/73 | 0/0 | 3/209 | 0
Pain (Any) (Skin and subcutaneous tissue disorders) | 265/331 | 0/0 | 221/301 | 0/0 | 286/322 | 0/0 | 62/79 | 0/0 | 73/87 | 0/0 | 139/164 | 0/0 | 161/173 | 0/0 | 761/787 | 0
Pain (Mild) (Skin and subcutaneous tissue disorders) | 254/323 | 0/0 | 199/290 | 0/0 | 263/306 | 0/0 | 58/76 | 0/0 | 68/83 | 0/0 | 125/156 | 0/0 | 150/165 | 0/0 | 672/721 | 0
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 48/206 | 0/0 | 63/210 | 0/0 | 75/190 | 0/0 | 13/53 | 0/0 | 26/59 | 0/0 | 57/111 | 0/0 | 60/112 | 0/0 | 360/467 | 0
Pain (Severe) (Skin and subcutaneous tissue disorders) | 3/178 | 0/0 | 16/187 | 0/0 | 5/139 | 0/0 | 1/48 | 0/0 | 4/44 | 0/0 | 10/86 | 0/0 | 4/75 | 0/0 | 38/238 | 0
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 61/214 | 0/0 | 65/211 | 0/0 | 79/194 | 0/0 | 15/54 | 0/0 | 24/57 | 0/0 | 54/112 | 0/0 | 56/109 | 0/0 | 375/499 | 0
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 57/212 | 0/0 | 61/208 | 0/0 | 73/189 | 0/0 | 13/54 | 0/0 | 23/57 | 0/0 | 51/110 | 0/0 | 51/106 | 0/0 | 333/466 | 0
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 4/179 | 0/0 | 7/182 | 0/0 | 4/140 | 0/0 | 2/47 | 0/0 | 3/43 | 0/0 | 3/81 | 0/0 | 7/77 | 0/0 | 44/238 | 0
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 3/180 | 0/0 | 8/185 | 0/0 | 4/139 | 0/0 | 1/47 | 0/0 | 2/41 | 0/0 | 8/84 | 0/0 | 4/77 | 0/0 | 37/237 | 0
Fatigue (General disorders) | 175/277 | 0/0 | 168/273 | 0/0 | 157/248 | 0/0 | 35/69 | 0/0 | 43/68 | 0/0 | 72/125 | 0/0 | 76/125 | 0/0 | 446/554 | 0
Headache (General disorders) | 136/252 | 0/0 | 141/259 | 0/0 | 162/246 | 0/0 | 23/60 | 0/0 | 32/64 | 0/0 | 64/118 | 0/0 | 76/123 | 0/0 | 429/527 | 0
Chills (General disorders) | 48/204 | 0/0 | 48/199 | 0/0 | 31/158 | 0/0 | 12/52 | 0/0 | 19/56 | 0/0 | 34/99 | 0/0 | 24/93 | 0/0 | 109/286 | 0
Rash (General disorders) | 32/194 | 0/0 | 25/192 | 0/0 | 21/148 | 0/0 | 12/51 | 0/0 | 9/49 | 0/0 | 31/95 | 0/0 | 11/81 | 0/0 | 53/249 | 0
Vomiting (General disorders) | 7/180 | 0/0 | 10/186 | 0/0 | 10/144 | 0/0 | 4/48 | 0/0 | 2/43 | 0/0 | 1/79 | 0/0 | 3/76 | 0/0 | 36/240 | 0
Decreased appetite (General disorders) | 43/202 | 0/0 | 45/207 | 0/0 | 42/166 | 0/0 | 11/52 | 0/0 | 17/54 | 0/0 | 22/93 | 0/0 | 22/89 | 0/0 | 202/363 | 0
New generalized muscle pain (General disorders) | 140/249 | 0/0 | 155/268 | 0/0 | 147/238 | 0/0 | 33/60 | 0/0 | 43/66 | 0/0 | 92/136 | 0/0 | 89/128 | 0/0 | 460/561 | 0
Aggravated generalized muscle pain (General disorders) | 70/215 | 0/0 | 84/225 | 0/0 | 75/188 | 0/0 | 14/51 | 0/0 | 24/58 | 0/0 | 40/101 | 0/0 | 33/95 | 0/0 | 207/370 | 0
New generalized joint pain (General disorders) | 48/197 | 0/0 | 65/216 | 0/0 | 52/165 | 0/0 | 10/53 | 0/0 | 13/53 | 0/0 | 21/91 | 0/0 | 31/93 | 0/0 | 128/307 | 0
Aggravated generalized joint pain (General disorders) | 51/205 | 0/0 | 44/206 | 0/0 | 43/168 | 0/0 | 7/51 | 0/0 | 11/49 | 0/0 | 16/91 | 0/0 | 22/88 | 0/0 | 77/269 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 12 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site injury (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury associated with device (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pallor (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 0 | 5 | 0 | 4 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 6 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 7 | 0 | 3 | 0 | 11 | 0
Nasopharyngitis (Infections and infestations) | 7 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 7 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fever Any (>=38 degrees C) (General disorders) | 14/181 | 0/0 | 11/185 | 0/0 | 2/137 | 0/0 | 1/48 | 0/0 | 2/43 | 0/0 | 2/79 | 0/0 | 2/75 | 0/0 | 16/221 | 0
Fever Mild (>=38 degrees C but <38.5 degrees C) (General disorders) | 7/179 | 0/0 | 2/180 | 0/0 | 2/137 | 0/0 | 0/47 | 0/0 | 1/42 | 0/0 | 2/79 | 0/0 | 2/75 | 0/0 | 9/214 | 0
Fever Moderate (>=38.5 degrees C but <39 degrees C) (General disorders) | 1/178 | 0/0 | 0/179 | 0/0 | 0/136 | 0/0 | 1/48 | 0/0 | 1/42 | 0/0 | 0/78 | 0/0 | 0/73 | 0/0 | 4/211 | 0
Fever Severe (>=39 degrees C but <=40 degrees C) (General disorders) | 0/177 | 0/0 | 0/179 | 0/0 | 0/136 | 0/0 | 0/47 | 0/0 | 0/41 | 0/0 | 0/78 | 0/0 | 0/73 | 0/0 | 3/210 | 0
Fever Potentially life threatening (>40 degrees C) (General disorders) | 8/180 | 0/0 | 9/184 | 0/0 | 0/136 | 0/0 | 0/47 | 0/0 | 0/41 | 0/0 | 0/78 | 0/0 | 0/73 | 0/0 | 1/208 | 0 — All reports of fever >40 degrees C in 13vPnC and 23vPS for Cohort 1 were confirmed as data entry errors.
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.